CLINICAL TRIAL: NCT01995552
Title: IdeNtifying High riSk Patients Post Myocardial Infarction With REduced Left Ventricular Function Using External Loop Recorders (INSPIRE-ELR Study)
Acronym: INSPIRE-ELR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version 3.0 , 22 Apr 2015; REF/2013/10/005823 (Other: Clinical Trial Registry - India)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Post MI Left Ventricular Dysfunction
Keywords: Post myocardial infarction patients with low EF.
MeSH Terms: interventions — Mucociliary Clearance; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External Loop Recorder (Other): This is a non-randomized study. All the patients will be enrolled will received the ELR system.
  Interventions: Device: External Loop Recorder

INTERVENTIONS:
Device: External Loop Recorder
  Other Names: NUVANT Mobile Cardiac Telemetry (MCT) system (CorventisTM); SEEQ™ External Cardiac Monitor (ECM) system (Medtronic, Inc., Minneapolis, MN)

SUMMARY:
The purpose of the INSPIRE-ELR study is to characterize arrhythmias in post MI low EF (≤35%) patients in the acute phase (at discharge from hospital after index MI) and chronic phase (at 8-10 weeks after index MI) and to correlate with patients at high risk of all-cause mortality or sudden cardiac death (SCD) at 1 year.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, interventional, non-randomized study enrolling post MI low left ventricular ejection fraction (LVEF ≤35%) patients prior to or at discharge from the hospital after index MI as defined in the inclusion criteria. Prior to initiating any study specific procedures, patients needs to provide his/her consent by signing and dating an informed consent form. Inclusion/Exclusion criteria will be evaluated and the patients' medical history and baseline information will be collected. Seven days ELR monitoring will be done at discharge and at chronic phase after index MI. At 6 and 9 months telephone follow-up will be done to evaluate the health status, if there will be no in-office visit planned. At 12 months there will be a scheduled in-office visit conducted to collect the health status. All the patients will be followed-up by telephone (health status) at study end (when the last patient completed the 12 month follow-up)

ELIGIBILITY:
Patients must meet all of the below criteria to be eligible for the study:

* Patients must provide written informed consent/data release consent to
* participate in the study.
* Acute Myocardial Infarction (STEMI or non-STEMI) documented within 10 days of onset, matching one of the following criteria:
* Acute ST segment elevation greater than or equal to 0.1 mv on ECG in 2 or more leads or new LBBB, with symptoms of ischemia
* In all other situations, including non ST segment elevation MI, at least one cardiac biomarker value [preferably cardiac troponin (cTn)] above the 99th percentile of a normal reference population (upper reference limit (URL)) AND with at least one of the following (1) new or presumed new ST-T changes (2) Symptoms or signs of Ischemia (3) Development of pathological Q waves in the ECG (4) Identification of an intracoronary thrombus by angiography
* LVEF less than or equal to 35 percent as measured by echocardiography Simpsons method, biplane one day before or on the day of hospital discharge

Exclusion Criteria

* Patients who cannot be discharged from the hospital within14 days after index Myocardial Infarction event
* Age less than 18 years
* Psychologically incapacitated
* Patient is pregnant, or is expecting to become pregnant during the course of the trial per Investigator discretion.
* Patients contraindicated for NUVANT system
* Comorbidities likely to limit survival to less than the minimal study duration (12 months)
* Participation in an investigational study with known or suspected cardiac effect expected to confound the results of this study (e.g. stem cell trials, stent trials, cardiac intervention trials, drug trials)
* Patients with an existing pacemaker or ICD implanted.
* Patients that are dialysis dependent at discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-02-20 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medanta - The Medicity, Gurgaon, Haryana, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled acute post MI patients with a reduced LVEF (≤35%) one day before or on the day of discharge from hospital after index MI. There is no control group in this study. The study was conducted in India and in multi specialty hospitals
Pre-assignment Details: The first patient was enrolled on April 29, 2014. Enrollment continued until the 250th patient was enrolled on January 31, 2016. out of 250, patients, there were 233 patients in the analysis cohort, with at least 72 hours of monitoring documented in the ELR device data or a clinically significant arrhythmia in the first 72 hours of monitoring.
Groups:
- External Loop Recorder (Single Arm): This is a non-randomized study. All the patients who were enrolled received the ELR system. (External Loop Recorder) After enrollment in the study the following visits are scheduled:
  * Baseline (day of discharge or one day before discharge after index MI). the main activities were Patient demographics, apply ELR, 12 lead ECG, LVEF etc.
  * Chronic phase follow-up visit: apply ELR, 12 lead ECG, LVEF etc. 6 and 9 months follow-up: Telephonic health status if patient is not seen.
  * 12-month follow-up visit: In office visit, health status questionnaire
  * Extended follow-up beyond 12 months: Telephonic health status at the study end (when the last patient completes the 12 months follow up).
Period: Overall Study
Arm/Group | External Loop Recorder (Single Arm)
Started (The study required to enroll 250 patients:) | 250 (There were 249 patients were included for Baseline cohort and 233 in analysis cohort)
Completed | 233 (There were 233 patients who were eligible for primary objective analysis)
Not Completed | 17
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 15
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The baseline cohort consists of 250 patients and the analysis cohort of 233. There were 17 patients excluded from the analysis because they were not fulfilling the required criteria of analysis as per the protocol.
Arm/Group | External Loop Recorder (Single Arm)
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 patient was excluded due to LVEF >35% which is the exclusion criteria
  Participants
    number analyzed (Participants) | 249
    <=18 years | 0
    Between 18 and 65 years | 192
    >=65 years | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: one patient was excluded due to LVEF>35 which is the exclusion criteria
  Participants
    number analyzed (Participants) | 249
    Female | 34
    Male | 215
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 250
Ejection Fraction [Mean (Standard Deviation); unit: % Ejection Fraction] — Population: The baseline cohort consists of 249 patients and the analysis cohort of 233.
  % Ejection Fraction
    number analyzed (Participants) | 249
    (all) | 31.7 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Study is to Assess Percent of Participants With Clinically Significant Arrhythmias on ELR Post MI
Description: Post MI mortality is higher in India than in the US and Western Europe. The hypothesis of the INSPIRE-ELR study was that occurrence of arrhythmias in the acute phase of MI will identify patients at highest risk and we evaluated the percentage clinical signification arrhythmias captured through the ELR post MI in acute phase
Time Frame: 7 days post discharge
Measure: Number (95% Confidence Interval); unit: percentage of analyzed population
Groups:
- External Loop Recorder (Single Arm): This is a non-randomized study. All the patients will be enrolled will received the ELR system.
Arm/Group | External Loop Recorder (Single Arm)
Number analyzed (Participants) | 233
percentage of analyzed population | 48.5 [42.2 to 54.9]

2. Secondary Outcome: Determine Percentage of Patients With Non-lethal Arrhythmias on ELR Post MI Have a Higher Risk of All-cause Mortality at 1 Year
Description: Analysis included all patients that completed the acute monitoring period. Based on the arrhythmias detected during the acute ELR monitoring period, patients were classified as "with arrhythmia" when during the ELR monitoring period there is any episode of ELR monitored events listed. All other patients are classified "without arrhythmia". Mortality rates after the monitoring period was estimated for both groups.
Time Frame: 12 Months
Population: There were total 28 deaths reported
Measure: Number (95% Confidence Interval); unit: percentage of Mortality
Groups:
- Acute Phase (With Arrhythmias): Patients were classified as "with significant arrhythmia" when during the ELR monitoring period and mortality was seen during 12 month follow-up.
- Acute Phase (Without Arrhythmias): Patients were classified as "without significant arrhythmia" when during the ELR monitoring period and mortality was seen during 12 month follow-up.
Arm/Group | Acute Phase (With Arrhythmias) | Acute Phase (Without Arrhythmias)
Number analyzed (Participants) | 113 | 120
percentage of Mortality | 19.6 [13.3 to 28.2] | 3.5 [1.3 to 9.0]

ADVERSE EVENTS:
Time Frame: All safety events were collected once the enrollment started and till the end of patient follow-ups during the period of 3 years
Description: As per the study protocol Deaths and Cardiovascular Related Serious Adverse Events were collected
Groups:
- External Loop Recorder (Single Arm): For this study, only Deaths and Cardiovascular Related Serious Adverse Events were collected. There were in total 28 deaths and 49 SAEs reported. No system or procedure related SAE were reported
Arm/Group | External Loop Recorder (Single Arm)
All-Cause Mortality (participants affected / at risk) | 28/249
Serious Adverse Events (participants affected / at risk) | 49/249
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | External Loop Recorder (Single Arm) (N=249)
Cardiac arrest (Cardiac disorders) | 4 (4) — Cardiac arrest
Acute left ventricular failure (Cardiac disorders) | 3 (3) — Acute left ventricular failure
Cardiac failure congestive (Cardiac disorders) | 3 (3) — Cardiac failure congestive
Coronary artery disease (Cardiac disorders) | 3 (3) — Coronary artery disease
Acute myocardial infarction (Cardiac disorders) | 2 (2) — Acute myocardial infarction
Ventricular tachyarrhythmia (Cardiac disorders) | 3 (3) — Ventricular tachyarrhythmia
Ventricular tachycardia (Cardiac disorders) | 3 (3) — Ventricular tachycardia
Angina pectoris (Cardiac disorders) | 1 (1) — Angina pectoris
Angina unstable (Cardiac disorders) | 1 (1) — Angina unstable
Atrial fibrillation (Cardiac disorders) | 1 (1) — Atrial fibrillation
Atrioventricular block complete (Cardiac disorders) | 1 (1) — Atrioventricular block complete
Cardiac failure (Cardiac disorders) | 1 (1) — Cardiac failure
Cardiac failure acute (Cardiac disorders) | 1 (1) — Cardiac failure acute
Left ventricular dysfunction (Cardiac disorders) | 1 (1) — Left ventricular dysfunction
Left ventricular failure (Cardiac disorders) | 1 (1) — Left ventricular failure
Death (General disorders) | 5 (5) — Death
Unevaluable event (General disorders) | 2 (2) — Unevaluable event
Chest discomfort (General disorders) | 1 (1) — Chest discomfort
Multi-organ failure (General disorders) | 1 (1) — Multi-organ failure
Sudden cardiac death (General disorders) | 1 (1) — Sudden cardiac death
Vascular stent restenosis (General disorders) | 1 (1) — Vascular stent restenosis
Cerebral infarction (Nervous system disorders) | 1 (1) — Cerebral infarction
Cerebrovascular disorder (Nervous system disorders) | 1 (1) — Cerebrovascular disorder
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dyspnoea
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute pulmonary oedema
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dyspnoea exertional
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypoxia
Aortic stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Aortic stenosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes